CLINICAL TRIAL: NCT06146374
Title: A Randomized, Double Blind, Placebo-Controlled, Multiple Ascending Dose, Phase 1 Study of SLV213 in Healthy Volunteers
Brief Title: Safety Study of SLV213 for the Treatment of COVID-19.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: DMID unanimously arrived at a recommendation to terminate the study after study met cohort halting criteria.
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-0027; 75N93022D00016
Record Dates: First submitted 2023-11-22; First posted 2023-11-24 (Actual); Results first posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2023-12-26

CONDITIONS: COVID-19
Keywords: Coronavirus; Covid-19; Double Blind; Healthy Volunteers; Multiple Ascending Dose; Phase 1; Placebo Controlled; Randomized; SLV213
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — N-pip-phenylalanine-homophenylalanine-vinyl sulfone phenyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 2 (Experimental): 600mg (6x 100mg capsules) of SLV213 (N=8) or placebo (N=4) administered orally every 12 hours for 7 days to healthy male and female participants 18-65 years of age.
  Interventions: Other: Placebo for SLV213; Drug: SLV213
- Group 3 (Experimental): 800mg (8x 100mg capsules) of SLV213 (N=8) or placebo (N=4) administered orally every 12 hours for 7 days to healthy male and female participants 18-65 years of age.
  Interventions: Other: Placebo for SLV213; Drug: SLV213
- Group1 (Experimental): 400mg (4x 100mg capsules) of SLV213 (N=8) or placebo (N=4) administered orally every 12 hours for 7 days to healthy male and female participants 18-65 years of age.
  Interventions: Other: Placebo for SLV213; Drug: SLV213

INTERVENTIONS:
Other: Placebo for SLV213 — Microcrystalline cellulose in a size 1 orange hard gelatin capsule.
Drug: SLV213 — SLV213 drug substance (K777) is 4-methylpiperazine-1-carboxylic acid, a vinyl sulfone cysteine protease inhibitor for the treatment of subjects infected with SARS-CoV-2. SLV213 is a white powder substance without excipients or stabilizer that will be packed into gelatin capsules which has been demonstrated to exhibit broad inhibitory properties against host cathepsins (e.g., Cathepsin L).

SUMMARY:
This Phase 1 double blind, placebo-controlled study will evaluate the safety, tolerability, and pharmacokinetics (PK) of multiple ascending doses (MAD) of SLV213 in healthy male and female participants, 18-65 years of age. This study will help to select the most likely suitable dose (e.g., at Maximum Tolerated Dose [MTD]) for the treatment of patients with COVID-19 in a pivotal study. This phase 1 double blind, placebo-controlled study will consist of three sequential cohorts of 12 participants each (8 SLV213 and 4 placebo), at doses of 400 mg every 12 hours (Q12h), 600 mg Q12h, and 800 mg Q12h administered orally (PO) for 7 days. After each cohort, a Safety Review Committee (SRC) will evaluate the safety of the regimen before proceeding to dose the next cohort. Randomization will occur into the respective cohorts as above. Upon meeting the Inclusion/Exclusion criteria, subjects will begin treatment with SLV213 or placebo per their assigned cohort. The primary objective is to evaluate the safety and tolerability of multiple ascending doses of SLV213 for 7 days in healthy participants.

DETAILED DESCRIPTION:
This Phase 1 double blind, placebo-controlled study will evaluate the safety, tolerability, and pharmacokinetics (PK) of multiple ascending doses (MAD) of SLV213 in healthy male and female participants, 18-65 years of age. This study will help to select the most likely suitable dose (e.g., at Maximum Tolerated Dose [MTD]) for the treatment of patients with COVID-19 in a pivotal study. This phase 1 double blind, placebo-controlled study will consist of three sequential cohorts of 12 participants each (8 SLV213 and 4 placebo), at doses of 400 mg every 12 hours (Q12h), 600 mg Q12h, and 800 mg Q12h administered orally (PO) for 7 days. After each cohort, a Safety Review Committee (SRC) will evaluate the safety of the regimen before proceeding to dose the next cohort. Randomization will occur into the respective cohorts as above. Upon meeting the Inclusion/Exclusion criteria, subjects will begin treatment with SLV213 or placebo per their assigned cohort. Participants will take their study drug in the fasted state prior to morning and evening meals and will remain as in-patient in the clinical trial unit (CTU) during all treatments and for approximately 48 hours (h) after the last dose for monitoring. After discharge from the CTU, participants will be monitored by CTU staff by telephone to assess for new adverse events and use of concomitant medication since the last visit or contact, approximately weekly for three weeks. Participants will be asked to return to the CTU for further assessment of moderate or severe adverse events (AEs) use of concomitant medications (ConMeds) since the last visit or contact, approximately weekly for three weeks. The primary objective is to evaluate the safety and tolerability of multiple ascending doses of SLV213 for 7 days in healthy participants. The secondary objective is to characterize the multiple dose PK of SLV213 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Able to understand and willing to be available for all study visits and comply with all study procedures including Lifestyle Considerations throughout the study.
3. Male and Female individuals, age 18-65 inclusive at time of enrollment.
4. Good general health by medical history (MH), physical examination (PE), and vital signs (VS), clinical laboratory tests and Electrocardiogram (ECG) within normal reference range.

   Note 1: Lab exceptions include: lab test values that are within Grade 1 range per the Toxicity Table (Appendix A) are acceptable if not considered to be clinically significant by the investigator (PI, sub-investigator, or authorized clinician), with the exception of liver function tests (LFT) (transaminases Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), alkaline phosphatase (AP), total and direct bilirubin, serum creatinine, estimated glomerular filtration rate (eGFR) per the CKD-EPI formula, and urine protein, which must be within the laboratory normal reference range.

   Note 2: Screening laboratory values that fall outside the laboratory normal reference ranges and the ranges are not listed within the Toxicity Table (Appendix A) (e.g., decrease activated partial thromboplastin time (aPTT)) that are deemed Not Clinically Significant by the PI will be acceptable.
5. Ability to take oral medication and be willing to adhere to the dosing regimen.
6. Women of childbearing potential1 must have practiced or use true abstinence2 or use at least one acceptable primary form of contraception3 for specified periods4 before, during and after dosing.

   Note 1: Not of childbearing potential - post-menopausal females (defined as having a history of amenorrhea for at least one year) or a documented status as being surgically sterile (hysterectomy, bilateral oophorectomy, salpingectomy, tubal ligation, or Essure placement with a history of documented radiological confirmation test at least 90 days after the procedure).

   Note 2: True abstinence is 100% of the time without sexual intercourse (the male's penis enters the female's vagina). Periodic abstinence [e.g., calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception).

   Note 3: Acceptable forms of primary contraception include a monogamous relationship with a vasectomized partner who has been vasectomized for 180 days or more before the participant receiving the study product, tubal ligation, non-hormonal, intrauterine device, (and if in a monogamous relationship with a male partner who uses a barrier method without spermicide) Note 4: Specified periods include at least 30 days prior to screening, during the period between screening and completion of dosing, and until at least 30 days following receipt of the last dose of study product.
7. Women of childbearing potential must have a negative serum Beta-human chorionic gonadotropin (HCG) pregnancy test at screening and a negative urine HCG pregnancy test at check-in (Day-1) within 24 hours before receiving the initial study product.
8. Male participants receiving the study product must use acceptable contraception and refrain from donating sperm from the day of first dose until 30 days after the last dose or be vasectomized.1 Note 1: Acceptable contraception includes abstinence from intercourse with a female of childbearing potential or use of a male condom without spermicide when engaging in any activity that allows for the passage of ejaculate to a female during the intervention period and for at least 30 days after ending study dosing, or surgical sterilization for 180 days or more.
9. Willing to avoid excessive physical exercise starting within 48 h prior to dosing and until discharge from the CTU on Day 9.
10. No history of acute febrile or infectious illness for at least 7 days prior to the administration of study drug.

Exclusion Criteria:

1. Pregnant or lactating.
2. History of any chronic disease that may increase risk to subject or interfere with endpoint assessment1:

   Note 1: With the exception of stable chronic medical conditions that do not require prescribed oral or injectable medications (e.g., Type 2 diabetes managed by diet only).
3. History of bradycardia, orthostatic hypotension or orthostatic tachycardia, Long COVID or history of dysautonomia.1 Note 1: Exception is sinus bradycardia (HR <60 bpm) in healthy participants (e.g., conditioned athletes) could be enrolled per investigator's clinical judgement.
4. Known history of a clinically significant food or drug allergy/hypersensitivity including known allergy/hypersensitivity to ingredients of the study drug or placebo.
5. Current seasonal allergies with ongoing symptoms for more than a week prior to dosing requiring glucocorticoids and/or frequent use of antihistamines for treatment.
6. History of any clinically significant disease or disorder, medical/surgical procedure, or trauma within 4 weeks prior to initiation of administration of study product(s).
7. History of any psychiatric condition that has required hospitalization in the last 12 months or subject is considered psychologically unstable by the investigator.
8. History of any substance use disorder or positive urine drug screening (UDS) test for illicit substances at Screening or Check-in (Day -1)1.

   Note 1: Any approved medical use of amphetamines, barbiturates, benzodiazepines, cannabis, tricyclic antidepressants and opiates will not be acceptable.
9. History of alcoholism or of binge1 or heavy alcohol drinking2 at any time in the 6 months before study product administration or positive urine alcohol test at Screening or Check-in (Day -1).

   Note 1: Binge drinking is defined as 5 or more drinks during a single occasion if male, or 4 or more if female.

   Note 2: Heavy drinking of alcohol is defined as consumption of more than 14 drinks of alcohol per week if male, or more than 7 drinks if female.
10. History of >/=10 pack-years of nicotine product1 consumption in the 5-year period before screening, or positive urine cotinine screen at Check-in (Day -1)2.

    Note 1: Nicotine products include cigarettes, e-cigarettes, pipe, cigar, chewing tobacco, nicotine patch.

    Note 2: Positive urine cotinine at Screening is allowed if negative at Check-in (Day -1).
11. Body mass index (BMI) </= 18 kg/m2 or >/= 32 kg/m2, or weight </= 100 lbs at Screening.
12. Prior exposure to SLV213 or K777 or K11777.
13. Use of any prohibited prescription or non-prescription medication within 14 days or 5 half-lives of the drug, whichever is longer, prior to study Check-in.
14. Use of any investigational drug product within 30 days or 5 half-lives (whichever is longer) before investigational product administration in this study.
15. Planned participation in a clinical research study that requires treatment with a study drug, blood draws or other invasive assessments during the study period (screening until final visit).
16. Blood or plasma donation of 500 mL within 3 months or more than 100 mL within 30 days before signing informed consent or planned donation prior to completion of this trial.
17. Positive viral serology tests for Human Immunodeficiency Virus (HIV), hepatitis B virus, or hepatitis C virus (HCV) at screening1 with one exception2:

    Note 1: Viral serology tests include HIV 1 and HIV 2 antibodies, Hepatitis B virus surface antigen (HBsAg), and HCV antibodies.

    Note 2: Do not exclude participants with HCV antibodies who have been successfully treated for Hepatitis C, do not take any treatment medications currently, do not use prohibited medications, have normal transaminases and are generally healthy.
18. Positive SARS-CoV-2 (COVID-19) molecular diagnostic test (Cue Care™ test) at Check-in (Day -1).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-04-09 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-07-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Altasciences Inc - Kansas City, Overland Park, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study population included healthy male and female adults, ages 18-65, inclusive, who met all eligibility criteria. Participants were enrolled at a single clinical trial unit between April 9, 2024 and June 10, 2024 and were recruited via IRB-approved strategies, including direct mailing, recruitment from an IRB-approved trial registry and local advertisements/flyers.
Groups:
- Cohort 1 - 400 mg SLV213: 400 mg (4 x 100 mg capsules) of SLV213 administered orally every 12 hours for 7 days to healthy male and female participants 18-65 years of age.
  SLV213: SLV213 drug substance (K777) is 4-methylpiperazine-1-carboxylic acid, a vinyl sulfone cysteine protease inhibitor for the treatment of participants infected with SARS-CoV-2. SLV213 is a white powder substance without excipients or stabilizer that was packed into gelatin capsules. SLV213 has been demonstrated to exhibit broad inhibitory properties against host cathepsins (e.g., Cathepsin L).
- Cohort 2 - 600 mg SLV213: 600 mg (6 x 100 mg capsules) of SLV213 administered orally every 12 hours for 7 days to healthy male and female participants 18-65 years of age.
  SLV213: SLV213 drug substance (K777) is 4-methylpiperazine-1-carboxylic acid, a vinyl sulfone cysteine protease inhibitor for the treatment of participants infected with SARS-CoV-2. SLV213 is a white powder substance without excipients or stabilizer that was packed into gelatin capsules. SLV213 has been demonstrated to exhibit broad inhibitory properties against host cathepsins (e.g., Cathepsin L).
  The study was terminated early due to halting criteria being met in Cohort 1, so this Cohort was not enrolled.
- Cohort 3 - 800 mg SLV213: 800 mg (8 x 100 mg capsules) of SLV213 administered orally every 12 hours for 7 days to healthy male and female participants 18-65 years of age.
  SLV213: SLV213 drug substance (K777) is 4-methylpiperazine-1-carboxylic acid, a vinyl sulfone cysteine protease inhibitor for the treatment of participants infected with SARS-CoV-2. SLV213 is a white powder substance without excipients or stabilizer that was packed into gelatin capsules. SLV213 has been demonstrated to exhibit broad inhibitory properties against host cathepsins (e.g., Cathepsin L).
  The study was terminated early due to halting criteria being met in Cohort 1, so this Cohort was not enrolled.
- Placebo: Placebo participants from Cohort 1. Placebo capsules were administered by the same route as active drug.
  Placebo for SLV213: Microcrystalline cellulose in a size 1 orange hard gelatin capsule.
Period: Overall Study
Arm/Group | Cohort 1 - 400 mg SLV213 | Cohort 2 - 600 mg SLV213 | Cohort 3 - 800 mg SLV213 | Placebo
Started | 11 | 0 | 0 | 5
Completed | 11 | 0 | 0 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1 - 400 mg SLV213: 400 mg (4 x 100 mg capsules) of SLV213 administered orally every 12 hours for 7 days to healthy male and female participants 18-65 years of age.
- Placebo: Placebo participants from Cohort 1. Placebo capsules were administered by the same route as active drug.
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - 400 mg SLV213 | Placebo | Total
Number analyzed (Participants) | 11 | 5 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (11.7) | 40.2 (14.1) | 45.1 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 1 | 7
  Male | 5 | 4 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 11 | 4 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 9 | 4 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.51 (3.33) | 27.70 (4.41) | 27.57 (3.55)

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Treatment-Emergent Adverse Events (TEAEs) by Maximum Severity
Description: The number of participants who experienced at least one unsolicited TEAE of any relatedness are summarized by the maximum severity recorded. A TEAE is defined as any untoward medical occurrence associated with the use of an intervention in humans, whether or not considered intervention-related. A TEAE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of medicinal (investigational) product. Any medical condition that was present at screening was considered a baseline finding and not reported as a TEAE. However, if the severity (i.e., grade) of any pre-existing medical condition increases, it was recorded as a TEAE.
Time Frame: Day 1 through Day 28
Population: The safety population includes all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 400 mg SLV213 | Placebo
Number analyzed (Participants) | 11 | 5
Participants
  None | 0 | 0
  Mild | 7 | 3
  Moderate | 4 | 2
  Severe | 0 | 0

2. Primary Outcome: Frequency of Related Treatment-Related TEAEs
Description: The number of participants who experienced at least one related unsolicited TEAE of any severity. A TEAE is defined as any untoward medical occurrence associated with the use of an intervention in humans, whether or not considered intervention-related. A TEAE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of medicinal (investigational) product. Any medical condition that was present at screening was considered a baseline finding and not reported as a TEAE. However, if the severity (i.e., grade) of any pre-existing medical condition increases, it was recorded as a TEAE. A TEAE is considered related if there is a reasonable possibility that the study intervention caused the TEAE, or there is a temporal relationship between the study intervention and event.
Time Frame: Day 1 through Day 28
Population: The safety population includes all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 400 mg SLV213 | Placebo
Number analyzed (Participants) | 11 | 5
Participants | 11 | 5

3. Primary Outcome: Frequency of Serious Adverse Events (SAEs)
Description: The number of participants who experienced at least one SAE throughout the course of the study. An AE is considered "serious" if, in the view of either the investigator or sponsor, it results in any of the following outcomes:
  * Death
  * A life-threatening adverse event
  * Inpatient hospitalization or prolongation of existing hospitalization
  * A persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, or
  * A congenital anomaly/birth defect.
Time Frame: Day 1 through Day 28
Population: The safety population includes all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 400 mg SLV213 | Placebo
Number analyzed (Participants) | 11 | 5
Participants | 0 | 0

4. Primary Outcome: Frequency of Laboratory AEs by Maximum Severity
Description: The number of participants who experienced at least one laboratory AE of any relatedness are summarized by the maximum severity recorded. Graded chemistry measurements include sodium, potassium, carbon dioxide, calcium, creatinine, blood urea nitrogen, fasting glucose, total protein, albumin, total bilirubin, alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, amylase, lipase, magnesium, and inorganic phosphorous. Graded hematology measurements include hemoglobin, platelets, white blood cells, neutrophils, lymphocytes, monocytes, basophils, and eosinophils. Graded coagulation measurements include prothrombin time and activated partial thromboplastin time. Graded urinalysis measurements include nitrite, urine protein, urine glucose, white blood cells, red blood cells, and bacteria. If a laboratory value met the threshold for an AE at baseline, subsequent safety laboratory results were only considered to be an AE if the grading worsened in severity.
Time Frame: Day 1 through Day 28
Population: The safety population includes all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 400 mg SLV213 | Placebo
Number analyzed (Participants) | 11 | 5
Participants
  None | 0 | 0
  Mild | 10 | 4
  Moderate | 0 | 1
  Severe | 1 | 0

5. Primary Outcome: Frequency of Treatment-Related Laboratory AEs
Description: The number of participants who experienced at least one related laboratory AE of any severity. Graded chemistry measurements include sodium, potassium, carbon dioxide, calcium, creatinine, blood urea nitrogen, fasting glucose, total protein, albumin, total bilirubin, alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, amylase, lipase, magnesium, and inorganic phosphorous. Graded hematology measurements include hemoglobin, platelets, white blood cells, neutrophils, lymphocytes, monocytes, basophils, and eosinophils. Graded coagulation measurements include prothrombin time and activated partial thromboplastin time. Graded urinalysis measurements include nitrite, urine protein, urine glucose, white blood cells, red blood cells, and bacteria. If a laboratory value met the threshold for an AE at baseline, subsequent safety laboratory results were only considered to be an AE if the grading worsened in severity.
Time Frame: Day 1 through Day 28
Population: The safety population includes all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 400 mg SLV213 | Placebo
Number analyzed (Participants) | 11 | 5
Participants | 11 | 5

6. Primary Outcome: Frequency of Electrocardiogram (ECG) AEs by Maximum Severity
Description: The number of participants who experienced at least one ECG AE of any relatedness are summarized by the maximum severity recorded. Graded ECG parameters include PR Internal and QTcF Interval.
Time Frame: Day 1 through Day 28
Population: The safety population includes all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 400 mg SLV213 | Placebo
Number analyzed (Participants) | 11 | 5
Participants
  None | 11 | 4
  Mild | 0 | 1
  Moderate | 0 | 0
  Severe | 0 | 0

7. Primary Outcome: Frequency of Treatment-Related ECG AEs
Description: The number of participants who experienced at least one related ECG AE of any severity. Graded ECG parameters include PR Internal and QTcF Interval.
Time Frame: Day 1 through Day 28
Population: The safety population includes all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 400 mg SLV213 | Placebo
Number analyzed (Participants) | 11 | 5
Participants | 0 | 1

8. Primary Outcome: Frequency of Early Terminations or Withdrawals Due to Treatment-Related TEAEs
Description: The number of participants who terminated early or were withdrawn due to a treatment-related TEAE. This outcome is used to assess the tolerability of the study treatment.
Time Frame: Day 1 through Day 28
Population: The safety population includes all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 400 mg SLV213 | Placebo
Number analyzed (Participants) | 11 | 5
Participants | 1 | 0

9. Primary Outcome: Frequency of TEAEs
Description: The number of participants who experienced at least one TEAE of any severity. This outcome is used to assess the tolerability of the study treatment.
Time Frame: Day 1 through Day 28
Population: The safety population includes all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 400 mg SLV213 | Placebo
Number analyzed (Participants) | 11 | 5
Participants | 11 | 5

10. Primary Outcome: Frequency of Grade 3 or Higher Laboratory AEs
Description: The number of participants who experienced at least one Grade 3 (severe) or higher laboratory AE. This outcome is used to assess the tolerability of the study treatment.
Time Frame: Day 1 through Day 28
Population: The safety population includes all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 400 mg SLV213 | Placebo
Number analyzed (Participants) | 11 | 5
Participants | 1 | 0

11. Primary Outcome: Frequency of Grade 3 or Higher Vital Signs AEs
Description: The number of participants who experienced at least one Grade 3 (severe) or higher vital signs AE. This outcome is used to assess the tolerability of the study treatment.
Time Frame: Day 1 through Day 28
Population: The safety population includes all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 400 mg SLV213 | Placebo
Number analyzed (Participants) | 11 | 5
Participants | 0 | 0

12. Primary Outcome: Frequency of Grade 3 or Higher ECG AEs
Description: The number of participants who experienced at least one Grade 3 (severe) or higher ECG AE. This outcome is used to assess the tolerability of the study treatment.
Time Frame: Day 1 through Day 28
Population: The safety population includes all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 400 mg SLV213 | Placebo
Number analyzed (Participants) | 11 | 5
Participants | 0 | 0

13. Primary Outcome: Frequency of Participants Who Received All Oral Medication Doses
Description: The number of participants who received all doses of study product. This outcome is used to assess the tolerability of the study treatment.
Time Frame: Day 1 through Day 28
Population: The safety population includes all participants who received at least one dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 - 400 mg SLV213 | Placebo
Number analyzed (Participants) | 11 | 5
Participants | 8 | 4

14. Secondary Outcome: Maximum Concentration (Cmax) of SLV213 in Plasma After Dose 1
Description: PK parameters were estimated from the SLV213 plasma concentration-time data after dose 1 using Phoenix WinNonlin Non-compartmental analysis.
Time Frame: 0 h through 12 h post dose 1
Population: The PK population includes all randomized participants, including replacement participants, who received at least one dose of study treatment and have at least one quantifiable post-dosing plasma concentration to use for the PK analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 - 400 mg SLV213
Number analyzed (Participants) | 11
ng/mL | 617.1 (65)

15. Secondary Outcome: Minimum Concentration (Cmin) of SLV213 in Plasma After Dose 1
Description: as for outcome 14
Time Frame: 0 h through 12 h post dose 1
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 - 400 mg SLV213
Number analyzed (Participants) | 11
ng/mL | 22.45 (43)

16. Secondary Outcome: Time of Maximum Concentration (Tmax) of SLV213 in Plasma After Dose 1
Description: as for outcome 14
Time Frame: 0 h through 12 h post dose 1
Population: as for outcome 14
Measure: Median (Full Range); unit: h
Arm/Group | Cohort 1 - 400 mg SLV213
Number analyzed (Participants) | 11
h | 2.00 [1.0 to 2.0]

17. Secondary Outcome: Time of Minimum Concentration (Tmin) of SLV213 in Plasma After Dose 1
Description: as for outcome 14
Time Frame: 0 h through 12 h post dose 1
Population: as for outcome 14
Measure: Median (Full Range); unit: h
Arm/Group | Cohort 1 - 400 mg SLV213
Number analyzed (Participants) | 11
h | 11.80 [8.0 to 11.9]

18. Secondary Outcome: Area Under the Concentration-Time Curve From 0 h (Pre-Dose) to Infinity (AUC0-inf) of SLV213 in Plasma After Dose 1
Description: PK parameters were estimated from the SLV213 plasma concentration-time data after dose 1 using Phoenix WinNonlin Non-compartmental analysis. AUC0-inf was estimated for parameters meeting the following lambda-z acceptance criteria: rsq_adjusted (adjusted r squared) >= 0.90 and includes at least 3 time points after Tmax.
Time Frame: 0 h through 12 h post dose 1
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Cohort 1 - 400 mg SLV213
Number analyzed (Participants) | 11
ng*h/mL | 2234.6 (65)

19. Secondary Outcome: Area Under the Concentration-Time Curve From 0 h (Pre-Dose) to 12 h (AUC0-12) of SLV213 in Plasma After Dose 1
Description: as for outcome 14
Time Frame: 0 h through 12 h post dose 1
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Cohort 1 - 400 mg SLV213
Number analyzed (Participants) | 11
ng*h/mL | 2172.4 (64)

20. Secondary Outcome: Area Under the Concentration-Time Curve From 0 h (Pre-Dose) to the Last Concentration Above the Lower Limit of Quantitation (AUC0-last) of SLV213 in Plasma After Dose 1
Description: as for outcome 14
Time Frame: 0 h through 12 h post dose 1
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Cohort 1 - 400 mg SLV213
Number analyzed (Participants) | 11
ng*h/mL | 2157.5 (66)

21. Secondary Outcome: Area Under the Concentration-Time Curve From 0 h (Pre-Dose) to the End of the Dosing Interval (AUC0-tau) of SLV213 in Plasma After Dose 1
Description: as for outcome 14
Time Frame: 0 h through 12 h post dose 1
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Cohort 1 - 400 mg SLV213
Number analyzed (Participants) | 11
ng*h/mL | 2172.4 (64)

22. Secondary Outcome: Terminal Half-Life (t1/2) of SLV213 in Plasma After Dose 1
Description: PK parameters were estimated from the SLV213 plasma concentration-time data after dose 1 using Phoenix WinNonlin Non-compartmental analysis. t1/2 was estimated for parameters meeting the following lambda-z acceptance criteria: rsq_adjusted (adjusted r squared) >= 0.90 and includes at least 3 time points after Tmax.
Time Frame: 0 h through 12 h post dose 1
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Cohort 1 - 400 mg SLV213
Number analyzed (Participants) | 11
h | 2.15 (22)

23. Secondary Outcome: Total Clearance (CLT) of SLV213 in Plasma After Dose 1
Description: PK parameters were estimated from the SLV213 plasma concentration-time data after dose 1 using Phoenix WinNonlin Non-compartmental analysis. CLT was estimated for parameters meeting the following lambda-z acceptance criteria: rsq_adjusted (adjusted r squared) >= 0.90 and includes at least 3 time points after Tmax.
Time Frame: 0 h through 12 h post dose 1
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Cohort 1 - 400 mg SLV213
Number analyzed (Participants) | 11
L/h | 179.0 (65)

24. Secondary Outcome: Terminal Phase Elimination Rate Constant (Ke) of SLV213 in Plasma After Dose 1
Description: PK parameters were estimated from the SLV213 plasma concentration-time data after dose 1 using Phoenix WinNonlin Non-compartmental analysis. Ke was estimated for parameters meeting the following lambda-z acceptance criteria: rsq_adjusted (adjusted r squared) >= 0.90 and includes at least 3 time points after Tmax.
Time Frame: 0 h through 12 h post dose 1
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | Cohort 1 - 400 mg SLV213
Number analyzed (Participants) | 11
1/h | 0.3220 (22)

25. Secondary Outcome: Volume of Distribution (Vd) of SLV213 in Plasma After Dose 1
Description: PK parameters were estimated from the SLV213 plasma concentration-time data after dose 1 using Phoenix WinNonlin Non-compartmental analysis. Vd was estimated for parameters meeting the following lambda-z acceptance criteria: rsq_adjusted (adjusted r squared) >= 0.90 and includes at least 3 time points after Tmax.
Time Frame: 0 h through 12 h post dose 1
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Cohort 1 - 400 mg SLV213
Number analyzed (Participants) | 11
L | 555.5 (63)

26. Secondary Outcome: Dose-normalized AUC0-Tau (AUC0-tau/Dose) of SLV213 in Plasma After Dose 1
Description: as for outcome 14
Time Frame: 0 h through 12 h post dose 1
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL/mg
Arm/Group | Cohort 1 - 400 mg SLV213
Number analyzed (Participants) | 11
ng*h/mL/mg | 5.428 (64)

27. Secondary Outcome: Dose-normalized Cmax (Cmax/Dose) of SLV213 in Plasma After Dose 1
Description: as for outcome 14
Time Frame: 0 h through 12 h post dose 1
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | Cohort 1 - 400 mg SLV213
Number analyzed (Participants) | 11
ng/mL/mg | 1.544 (65)

28. Secondary Outcome: Cmax at Steady State (Cmax,ss) of SLV213 in Plasma After Dose 14
Description: PK parameters were estimated from the SLV213 plasma concentration-time data after dose 14 (the last dose) using Phoenix WinNonlin Non-compartmental analysis. The estimate assumes steady state has been achieved.
Time Frame: 0 h through 48 h post dose 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 - 400 mg SLV213
Number analyzed (Participants) | 8
ng/mL | 419.0 (58)

29. Secondary Outcome: Cmin at Steady State (Cmin,ss) of SLV213 in Plasma After Dose 14
Description: as for outcome 28
Time Frame: 0 h through 48 h post dose 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 - 400 mg SLV213
Number analyzed (Participants) | 8
ng/mL | 23.66 (47)

30. Secondary Outcome: Average Concentration During the Dosing Interval (Cavg) of SLV213 in Plasma After Dose 14
Description: as for outcome 28
Time Frame: 0 h through 48 h post dose 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1 - 400 mg SLV213
Number analyzed (Participants) | 8
ng/mL | 135.2 (58)

31. Secondary Outcome: Tmax at Steady State (Tmax,ss) of SLV213 in Plasma After Dose 14
Description: as for outcome 28
Time Frame: 0 h through 48 h post dose 14
Population: as for outcome 14
Measure: Median (Full Range); unit: h
Arm/Group | Cohort 1 - 400 mg SLV213
Number analyzed (Participants) | 8
h | 2.00 [1.0 to 2.1]

32. Secondary Outcome: Tmin at Steady State (Tmin,ss) of SLV213 in Plasma After Dose 14
Description: as for outcome 28
Time Frame: 0 h through 48 h post dose 14
Population: as for outcome 14
Measure: Median (Full Range); unit: h
Arm/Group | Cohort 1 - 400 mg SLV213
Number analyzed (Participants) | 8
h | 12.05 [12.0 to 12.2]

33. Secondary Outcome: Area Under the Concentration-Time Curve From 0 h (Pre-Dose) to 48 h at Steady State (AUC0-48,ss) of SLV213 in Plasma After Dose 14
Description: as for outcome 28
Time Frame: 0 h through 48 h post dose 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Cohort 1 - 400 mg SLV213
Number analyzed (Participants) | 8
ng*h/mL | 1734.6 (56)

34. Secondary Outcome: AUC0-tau at Steady State (AUC0-tau,ss) of SLV213 in Plasma After Dose 14
Description: as for outcome 28
Time Frame: 0 h through 48 h post dose 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Cohort 1 - 400 mg SLV213
Number analyzed (Participants) | 8
ng*h/mL | 1624.4 (58)

35. Secondary Outcome: t1/2 of SLV213 in Plasma After Dose 14
Description: PK parameters were estimated from the SLV213 plasma concentration-time data after dose 14 (the last dose) using Phoenix WinNonlin Non-compartmental analysis. t1/2 was estimated for parameters meeting the following lambda-z acceptance criteria: rsq_adjusted (adjusted r squared) >= 0.90 and includes at least 3 time points after Tmax.
Time Frame: 0 h through 48 h post dose 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | Cohort 1 - 400 mg SLV213
Number analyzed (Participants) | 8
h | 3.05 (20)

36. Secondary Outcome: CLT at Steady State (CLT,ss) of SLV213 in Plasma After Dose 14
Description: as for outcome 28
Time Frame: 0 h through 48 h post dose 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Cohort 1 - 400 mg SLV213
Number analyzed (Participants) | 8
L/h | 246.1 (58)

37. Secondary Outcome: Vd at Steady State (Vd,ss) of SLV213 in Plasma After Dose 14
Description: as for outcome 28
Time Frame: 0 h through 48 h post dose 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L
Arm/Group | Cohort 1 - 400 mg SLV213
Number analyzed (Participants) | 8
L | 1079.1 (73)

38. Secondary Outcome: Dose-Normalized AUC0-tau,ss (AUC0-tau,ss/Dose) of SLV213 in Plasma After Dose 14
Description: as for outcome 28
Time Frame: 0 h through 48 h post dose 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL/mg
Arm/Group | Cohort 1 - 400 mg SLV213
Number analyzed (Participants) | 8
ng*h/mL/mg | 4.061 (58)

39. Secondary Outcome: Dose-Normalized Cmax,ss (Cmax,ss/Dose) of SLV213 in Plasma After Dose 14
Description: as for outcome 28
Time Frame: 0 h through 48 h post dose 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Arm/Group | Cohort 1 - 400 mg SLV213
Number analyzed (Participants) | 8
ng/mL/mg | 1.047 (58)

40. Secondary Outcome: Linearity Index of SLV213 in Plasma
Description: Linearity index is estimated as AUC0-tau,ss (Dose 14)/AUC0-inf (Dose 1). PK parameters were estimated from the SLV213 plasma concentration-time data after dose 1 and dose 14 (the last dose) using Phoenix WinNonlin Non-compartmental analysis.
Time Frame: 0 h through 12 h post dose 1, 0 h through 48 h post dose 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Cohort 1 - 400 mg SLV213
Number analyzed (Participants) | 8
ratio | 0.625 (40)

41. Secondary Outcome: Accumulation Ratio for AUC (RAUC) of SLV213 in Plasma
Description: RAUC is estimated as AUC0-tau,ss (Dose 14)/AUC0-tau (Dose 1). PK parameters were estimated from the SLV213 plasma concentration-time data after dose 1 and dose 14 (the last dose) using Phoenix WinNonlin Non-compartmental analysis.
Time Frame: 0 h through 12 h post dose 1, 0 h through 48 h post dose 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Cohort 1 - 400 mg SLV213
Number analyzed (Participants) | 8
ratio | 0.641 (40)

42. Secondary Outcome: Accumulation Ratio for Cmax (RCmax) of SLV213 in Plasma
Description: RCmax is estimated as Cmax,ss (Dose 14)/Cmax (Dose 1). PK parameters were estimated from the SLV213 plasma concentration-time data after dose 1 and dose 14 (the last dose) using Phoenix WinNonlin Non-compartmental analysis.
Time Frame: 0 h through 12 h post dose 1, 0 h through 48 h post dose 14
Population: 0 h through 12 h post dose 1, 0 h through 48 h post dose 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Cohort 1 - 400 mg SLV213
Number analyzed (Participants) | 8
ratio | 0.598 (47)

ADVERSE EVENTS:
Time Frame: All TEAEs were documented from time of starting drug administration through the time of the last assessment (e.g., Day 8 for clinical safety labs and ECGs) or Final Visit (Day 28 +/- 2 days).
Description: Any systemic medical condition, vital sign and ECG measurement, and clinical safety lab test value that was present on Day 1 prior to dosing was considered a baseline findings. If the condition increases in severity or frequency after study product administration, it was reported as a TEAE.
Arm/Group | Cohort 1 - 400 mg SLV213 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/5
Other Adverse Events (participants affected / at risk) | 11/11 | 5/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 - 400 mg SLV213 (N=11) | Placebo (N=5)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Eructation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (2)
Drug hypersensitivity (Immune system disorders) | 2 (2) | 0 (0) — The study was terminated early due to reporting of this event in two participants.
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood pressure diastolic increased (Investigations) | 1 (1) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 1 (3)
Electrocardiogram PR prolongation (Investigations) | 0 (0) | 1 (1)
Heart rate decreased (Investigations) | 3 (8) | 2 (5)
Orthostatic heart rate response increased (Investigations) | 7 (23) | 2 (9)
Respiratory rate increased (Investigations) | 11 (47) | 4 (12)
Dizziness (Nervous system disorders) | 10 (14) | 4 (7)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Taste disorder (Nervous system disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (3)
Amylase increased (Investigations) | 1 (4) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Blood calcium decreased (Investigations) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 3 (3) | 0 (0)
Blood phosphate decrease decreased (Investigations) | 1 (1) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 1 (1)
Blood sodium increased (Investigations) | 1 (2) | 0 (0)
Glucose urine present (Investigations) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 10 (28) | 5 (17)
Lymphocyte count decreased (Investigations) | 2 (2) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1)
Protein total decreased (Investigations) | 1 (2) | 0 (0)
Protein urine present (Investigations) | 1 (1) | 0 (0)
Prothrombin time prolonged (Investigations) | 2 (2) | 0 (0)
Red blood cells urine positive (Investigations) | 1 (2) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 1 (1)
White blood cells urine positive (Investigations) | 2 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol (2024-03-27): https://cdn.clinicaltrials.gov/large-docs/74/NCT06146374/Prot_001.pdf
  • Statistical Analysis Plan (2024-11-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT06146374/SAP_002.pdf
  • Informed Consent Form (2024-03-11): https://cdn.clinicaltrials.gov/large-docs/74/NCT06146374/ICF_000.pdf